CLINICAL TRIAL: NCT06095219
Title: MRI-based 3D Hip Labrum and Cartilage Morphology in Patients With Hip Deformities Compared to Asymptomatic Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 5273; 320030_205091 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hip Disease
Keywords: Hip dysplasia; Acetabular protrusion; Deep hip; Acetabular retroversion
MeSH Terms: conditions — Hip Dislocation | interventions — Magnetic Resonance Spectroscopy; Contrast Media

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Asymptomatic volunteers: Healthy individuals without history of hip pain or problems willing to undergo MRI of the hip.
  Interventions: Other: Non- contrast Magnetic Resonance Imaging (MRI) of the hip
- Hip Dysplasia: This group is defined according to the following radiographic parameter: lateral center edge angle (LCE) < 23°. The data was obtained from a retrospective study.
  Interventions: Other: Magnetic Resonance Imaging (MRI) of the hip with intra-articular contrast agent
- cam Deformity: This group is defined according to the following radiographic parameter: alpha angle > 60°. The data was obtained from a retrospective study.
  Interventions: Other: Magnetic Resonance Imaging (MRI) of the hip with intra-articular contrast agent
- Acetabular retroversion: This group is defined according to the following radiographic parameters:positive posterior- wall- sign, positive ischial spine sign, and positive cross- over- sign. The data was obtained from a retrospective study.
  Interventions: Other: Magnetic Resonance Imaging (MRI) of the hip with intra-articular contrast agent
- Acetabular protrusion: This group is defined according to the following radiographic parameter: positive protrusion sign. The data was obtained from a retrospective study.
  Interventions: Other: Magnetic Resonance Imaging (MRI) of the hip with intra-articular contrast agent
- Deep hip: This group is defined according to the following radiographic parameter: LCE angle > 39°. The data was obtained from a retrospective study.
  Interventions: Other: Magnetic Resonance Imaging (MRI) of the hip with intra-articular contrast agent

INTERVENTIONS:
Other: Non- contrast Magnetic Resonance Imaging (MRI) of the hip — Asymptomatic volunteers will undergo a non-contrast MRI of the hip at 3 Tesla. Following this, MRI images will be automatically segmented utilizing a validated artificial intelligence based algorithm to calculate 3D outcome parameters.
  Groups: Asymptomatic volunteers
Other: Magnetic Resonance Imaging (MRI) of the hip with intra-articular contrast agent — The data was derived from a retrospective study involving patients at Inselspital's outpatient clinic who underwent 3 Tesla hip MRI scans with intra-articular contrast agent. A validated artificial intelligence based algorithm was utilized for automated segmentation and the calculation of 3D outcome parameters.
  Groups: Acetabular protrusion; Acetabular retroversion; Deep hip; Hip Dysplasia; cam Deformity

SUMMARY:
In this study, the investigators seek to describe the normal 3D hip joint morphology in asymptomatic volunteers and compare it to various hip joint deformities. Asymptomatic volunteers will be asked to undergo a non-contrast MRI of the hip at 3 Tesla, utilizing a high-resolution morphologic 3D sequence (3D T2 DESS) that enables the segmentation of labrum and cartilage. 3D morphological parameters of the asymptomatic group will subsequently be compared with the 3D morphological parameters of patients with hip deformities, which were collected as part of a previous retrospective study.

DETAILED DESCRIPTION:
Hip deformities can cause hip pain and early onset osteoarthritis in young individuals.

Correcting these deformities typically involves planning with X-rays and MRI images, which offer a limited view of the hip joint's 3D structure. A comprehensive 3D analysis of hip structures, including cartilage, and labrum, would enhance diagnosis and surgery planning. However, 3D hip morphology hasn't been adequately described for distinguishing deformities.

The aim of this study is to describe normal 3D hip joint morphology in healthy participants and compare it to various hip joint deformities (Dysplasia, acetabular protrusion, retroversion, deep hip, and cam deformity).

Asymptomatic volunteers will undergo a non-contrast MRI of the hip at 3 Tesla using high-resolution morphologic 3D sequence (3D T2 DESS), which allows segmentation of labrum and cartilage.

The 3D morphological parameters of the asymptomatic group will then be compared with those of patients with hip deformities, data sourced from a retrospective study that included 100 patients from the outpatient clinic. These patients underwent direct MR arthrography at 3 Tesla in accordance with the institutional routine protocol at the Department of Diagnostic, Interventional, and Pediatric Radiology at Inselspital.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years.
* Signed an informed consent form.
* History free of significant hip pain, with no history of juvenile hip disease, traumatic injuries, inflammatory conditions, or tumors affecting the hip.
* Normal clinical examination of the hip.

Exclusion Criteria:

Individuals who are not considered suitable for MRI (Magnetic Resonance Imaging) for the following reasons:

* Potential pregnancy
* Presence of metal fragments in the eye or elsewhere in the body
* Presence of implants and metallic foreign bodies, such as a pacemaker, heart valve, cerebrospinal fluid shunt, insulin pump, nerve stimulator, or cochlear implant
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be publicly advertised in the Bern area. Interested individuals can contact by phone or electronically. Study information will be provided, and appointments will be scheduled for clinical exams and, if deemed necessary based on eligibility criteria, an MRI. Informed consent interviews will be conducted by investigators. MRI procedures will follow, without the use of contrast medium or ionizing radiation. Data for comparison will be obtained from a retrospective study involving 100 patients with hip deformities from the outpatient clinic who underwent direct MR arthrography at 3 Tesla.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cartilage Surface Area | Within 12 Months after MRI
  Difference in hip cartilage surface area (both absolute - mm² and relative - %) between healthy volunteers and patients with hip deformities.
Cartilage Thickness | Within 12 Months after MRI
  Difference in hip cartilage thickness (mm) between healthy volunteers and patients with hip deformities
Cartilage Orientation | Within 12 Months after MRI
  Difference in hip cartilage orientation, measured in inclination (°) and anteversion (°), between healthy volunteers and patients with hip deformities.
Cartilage Volume | Within 12 Months after MRI
  Difference in hip cartilage volume (mm³) between healthy volunteers and patients with hip deformities.
Labrum Length | Within 12 Months after MRI
  Difference in labrum length (mm) between healthy subjects and patients with hip deformities.
Labrum Area | Within 12 Months after MRI
  Difference in hip labrum surface area (both absolute - mm² and relative - %) between healthy volunteers and patients with hip deformities.
Labrum Volume | Within 12 Months after MRI
  Difference in hip labrum volume (mm³) between healthy volunteers and patients with hip deformities.

SECONDARY OUTCOMES:
iHOT 12 Questionnaire | ca. 5 minutes before MRI
  The iHOT-12 is a validated questionnaire for young, active individuals with early hip disease. It covers four domains: symptoms and limitations, sports and recreation, job concerns, and social/emotional aspects. Responses are marked on a 100-mm scale, with the total score as a simple mean ranging from 0 to 100, where 100 represents the best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Simon D. Steppacher, Dr., Principal Investigator — University Hospital of Bern (Inselspital)
Locations (1):
- University Hospital of Bern (Inselspital), Bern, Switzerland